CLINICAL TRIAL: NCT06378658
Title: A Phase 1, Open Label, Randomized, Crossover Study to Investigate the Effect of Food and Effect of an Acid Reducing Agent on the Pharmacokinetics of BAY 2927088 in Healthy Participants
Brief Title: A Study to Learn About How Food and Esomeprazole Affect the Level of BAY2927088 in the Blood When Taken Together in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 22253
Record Dates: First submitted 2024-03-19; First posted 2024-04-22 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Advanced Non-small Cell Lung Cancer; EGFR Mutation; HER2 Mutation; Healthy Volunteers
Keywords: HER2; EGFR; NSCLC
MeSH Terms: interventions — Esomeprazole; Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Intervention A - Intervention B - Intervention C (Experimental): Intervention A: BAY2927088 is administered under fasted status. Intervention B: BAY2927088 is administered under fed status (light low-fat meal).
  Intervention C: BAY2927088 is administered under fed status (high fat, high calorie meal).
  Each participant will subsequently undergo a fourth intervention period that includes dosing with BAY2927088 and esomeprazole.
  Interventions: Drug: BAY2927088; Drug: Esomeprazole; Other: Food
- Intervention B - Intervention C- Intervention A (Experimental): Intervention A: BAY2927088 is administered under fasted status. Intervention B: BAY2927088 is administered under fed status (light low-fat meal).
  Intervention C: BAY2927088 is administered under fed status (high fat, high calorie meal).
  Each participant will subsequently undergo a fourth intervention period that includes dosing with BAY2927088 and esomeprazole.
  Interventions: Drug: BAY2927088; Drug: Esomeprazole; Other: Food
- Intervention C - Intervention A - Intervention B (Experimental): Intervention A: BAY2927088 is administered under fasted status. Intervention B: BAY2927088 is administered under fed status (light low-fat meal).
  Intervention C: BAY2927088 is administered under fed status (high fat, high calorie meal).
  Each participant will subsequently undergo a fourth intervention period that includes dosing with BAY2927088 and esomeprazole.
  Interventions: Drug: BAY2927088; Drug: Esomeprazole; Other: Food

INTERVENTIONS:
Drug: BAY2927088 — Oral administration
Drug: Esomeprazole — Oral administration
Other: Food — light low-fat meal or high fat, high calorie meal

SUMMARY:
Researchers are looking for a better way to treat people who have advanced non-small cell lung cancer (NSCLC) with specific genetic changes called epidermal growth factor receptor (EGFR) and human epidermal growth factor receptor 2 (HER2) mutations.

Advanced NSCLC refers to a type of lung cancer that has spread from the lungs to nearby tissues or other body parts. People with advanced NSCLC may have changes in certain proteins, like EGFR and HER2, that cause uncontrolled cell growth and increased spread of cancer.

In this study, participants will be healthy and will not benefit from taking the study treatment, BAY2927088. However, the study will provide information about how to test BAY2927088 in future studies with people who have advanced NSCLC with EGFR or HER2 mutations.

BAY2927088 is under development for the treatment of advanced NSCLC with EGFR or HER2 mutations. It is expected to work against these changed proteins, which might slow down the spread of cancer.

The absorption of BAY2927088 into the blood is dependent on the amount of acid present in the stomach. Esomeprazole is a medicine which is used in the treatment of heartburn and excessive acid in the stomach. Both food and esomeprazole may change the amount of acid present in the stomach.

The main purpose of this study is to find out how food and esomeprazole may affect the absorption of BAY2927088 into the blood of healthy participants. For this, researchers will measure the levels of BAY2927088 in participants' blood when it is given with or without food as well as with or without esomeprazole. Researchers will then calculate the following:

* Area under the curve (AUC): a measure of the total amount of BAY2927088 in participants' blood over time
* Maximum observed concentration (Cmax): the highest amount of BAY2927088 in participants' blood

The study will have 4 treatment periods:

- Periods 1 to 3 (Day 1 to Day 9): All participants will take BAY2927088 with a low-fat meal, with a high-fat meal, and on an empty stomach, but in a different order, over the 3 study periods. Each period will last for 3 days and BAY2927088 will be given on the first day of each period.

On Day 9, participants will take esomeprazole on an empty stomach.

- Period 4 (Day 10 to Day 14): On Days 10 and 11, participants will take esomeprazole on an empty stomach. On Day 12, participants will take esomeprazole on an empty stomach. After 1 and a half hours, participants will take low-fat meal and BAY2927088.

On Day 13, participants will take esomeprazole on an empty stomach.

Participants will be in this study for about 8 weeks with 3 visits to the study clinic.

Participants will visit the study clinic:

* at least once, 2 to 28 days before the treatment starts, to confirm they can take part in this study
* once on the day before the treatment starts and will stay in the clinic until Day 14 of the treatment
* once, 7 to 10 days after last dose of BAY2927088, for a health check-up

During the study, the doctors and their study team will:

* do physical examinations
* collect blood samples from the participants to measure the levels of BAY2927088
* check participants' health by performing tests, such as blood and urine tests, and checking heart health using an electrocardiogram (ECG)
* ask the participants questions about how they are feeling and what adverse events they are having An adverse event is any medical problem that a participant has during a study. The study doctors keep track of all adverse events, irrespective of whether they think it is related or not to the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent as described in protocol which includes compliance with the requirements and restrictions listed in the informed consent form (ICF), and in this protocol.
* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by the investigator or medically qualified designee based on medical evaluation including medical history, laboratory tests, physical, and cardiac examination.
* Participant is a nonsmoker who has not used tobacco- or nicotine- containing products (e.g., nicotine patch) for at least 6 months before administration of the first study intervention.
* Body mass index (BMI) within the range 18.0 to 30 kg/m^2 (inclusive) at screening, with bodyweight above/equal to 50 kg.
* Female, of non-childbearing potential only

  * Females must not be pregnant or breastfeeding and must be documented as a woman of nonchildbearing potential. A negative pregnancy test is required.
  * Male study participants of reproductive potential must agree to use adequate contraception when sexually active.
* From signing of the ICF until at least 3 months after the last dose of study intervention, and refrain from sperm donation during study intervention and for 3 months after the last dose of study intervention.
* Participant must be willing to comply with dietary and fluid requirements during the study period (including abstaining from alcohol use).

Exclusion Criteria:

* Existing relevant diseases of vital organs (e.g., liver diseases, heart diseases, gastrointestinal diseases, interstitial lung disease, renal diseases), central nervous system (for example seizures) or other organs (e.g., diabetes mellitus).
* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination, and effects of the study intervention will not be normal.
* Febrile illness within 4 weeks prior to admission to the clinic.
* Any relevant diseases within 4 weeks prior to the first study intervention administration as judged by the investigator.
* A medical history of risk factors for Torsades de pointes (e.g., family history of long QT syndrome) or other clinically significant arrhythmias as judged by the investigator.
* Known severe allergies, allergies requiring therapy with corticosteroids, significant non-allergic drug reactions, or (multiple) drug allergies (excluding seasonal allergies such as non-severe hay fever that are asymptomatic and untreated during the time of study conduct).
* Known history of hypersensitivity (or known allergic reaction) to BAY 2927088-related compounds, or any components of the formulation, or esomeprazole.
* History of known or suspected malignant tumors.
* Participants with any type of ongoing psychiatric disorder, especially any mood disorders including medical history with suicidal ideation and/or suicide attempts, which may disable the participant to consent.
* Loss or donation (incl. plasmapheresis) of more than 100 mL of whole blood within 4 weeks or 500 mL of whole blood within 3 months before the first study intervention administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2024-03-29 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Cmax for BAY2927088 in plasma | Pre-dose on Day 1, 4, 7 and 12. Multiple post-dose time points on Day 1-2, Day 4-5, Day 7-8 and Day 12-13; one timepoint on Day 3, Day 6, Day 9 and Day 14
AUC for BAY2927088 in plasma | Pre-dose on Day 1, 4, 7 and 12. Multiple post-dose time points on Day 1-2, Day 4-5, Day 7-8 and Day 12-13; one timepoint on Day 3, Day 6, Day 9 and Day 14

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Up to 7 days after the last dose of BAY2927088

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel Baltimore - Early Phase Clinical Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here for access to information about Bayer's transparency standards and Bayer studies. — https://clinicaltrials.bayer.com/study/22253